CLINICAL TRIAL: NCT07200375
Title: Evaluating Effectiveness and Safety of Glofitamab Based Second-Line Therapy in Chinese Adult Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma: A Prospective, Observational, Multicenter, Cohort Study
Brief Title: An Observational Study of Glofitamab in Chinese Adult Participants With 2L Diffuse Large B-Cell Lymphoma
Acronym: GlofitReal
Status: Recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML45172
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — glofitamab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Glofitamab treatment: Participants will be enrolled into the study either prior to initiation of glofitamab therapy or within 90 days of starting glofitamab therapy.
  Interventions: Drug: Glofitamab

INTERVENTIONS:
Drug: Glofitamab — Participants will receive glofitamab as part of a cancer-treatment regimen in a real-world setting. No intervention will be administered by study investigators.

SUMMARY:
This study will investigate how well glofitamab-based therapy works and how safe it is in Chinese adult participants with relapsed or refractory diffuse large B-cell lymphoma (R/R DLBCL).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed R/R DLBCL after one line of systemic therapy
* Will be treated with Glofit-based regimen (known as being recommended and having the intention to be treated with Glofitamab at the time of signing ICF) or have initiated Glofit-based regimen treatment within three months (90 days) prior to enrollment

Exclusion Criteria:

* Participants who currently participate in or plan to participate in any interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Chinese participants with R/R DLBCL who will be treated with a glofitamab-based regimen either after enrollment into the study or within 90 days prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2029-09-29 (Estimated); Study Completion 2029-09-29 (Estimated)

PRIMARY OUTCOMES:
real-world Progression-Free Survival (rwPFS) | Up to approximately 4 years

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | Up to approximately 4 years
  CRR is defined as the proportion of participants whose best overall response (BOR) is a complete response (CR) on positron emission tomography/computed tomography (PET/CT) or CT during the study assessed by the investigator according to 2014 Lugano Response Criteria for Malignant Lymphoma
Overall Response Rate (ORR) | Up to approximately 4 years
  ORR is defined as the proportion of patients whose BOR is a CR or a partial response (PR) during the study assessed by the investigator according to 2014 Lugano Response Criteria for Malignant Lymphoma
Disease Control Rate (DCR) | Up to approximately 4 years
  DCR is defined as the proportion of patients achieving CR, PR or stable disease (SD) during the study assessed by the investigator according to 2014 Lugano Response Criteria for Malignant Lymphoma
Duration of Response (DoR) | Up to approximately 4 years
  DoR is defined as the time interval from the first occurrence of a documented objective response (CR or PR) to disease progression or death from any cause, whichever occurs first assessed by the investigator according to 2014 Lugano Response Criteria for Malignant Lymphoma
Duration of Complete Response (DoCR) | Up to approximately 4 years
  DoCR is defined as the time interval from the first occurrence of a documented CR to disease progression or death from any cause, whichever occurs first
Overall Survival (OS) | Up to approximately 4 years
  OS is defined as the time from treatment start of the Glofit-based regimen until the date of death from any cause
Event-Free Survival (EFS) | Up to approximately 4 years
  EFS is defined as the time from treatment start of the Glofit-based regimen to any treatment failure including disease progression, relapse, initiation of new antilymphoma therapy (NALT), or death from any cause, which occurs first, as determined by the investigator assessment according to 2014 Lugano Response Criteria for Malignant Lymphoma
Time to Next Treatment (TTNT) | Up to approximately 4 years
  TTNT is defined as the time from treatment start of the Glofit-based regimen to the initiation of next-line treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- China (12):
  - Chinese Academy of Medical Sciences Hematology Hospital;Lymphoma Diagnosis and Treatment Center, Tianjin, Tianjin Municipality
  - Peking University Third Hospital, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - Guangdong Provincial People's Hospital, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shandong Cancer Hospital, Jinan
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Xiehe Hospital, Tongji Medical College Huazhong University of Science & Technology, Wuhan
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No